CLINICAL TRIAL: NCT02119793
Title: A Multicenter, Extension Clinical Study to Evaluate the Long-term Efficacy and Safety of Repeat Treatment of YVOIRE Contour Injected Into the Anteromedial Malar Region in Subjects Who Have Completed the LG-HACL014 Study
Brief Title: Extension Clinical Study to Evaluate the Long-term Efficacy and Safety of Repeat Treatment of YVOIRE Contour Injected Into the Anteromedial Malar Region in Subjects Who Have Completed the LG-HACL014 Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-HACL015
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Normal, Healthy Adults With Moderate, Severe, or Very Severe Volume Loss of Anteromedial Malar Region Who Have Completed the LG-HACL014 Study

ARMS (1):
- YVOIRE contour (Experimental)
  Interventions: Device: YVOIRE contour

INTERVENTIONS:
Device: YVOIRE contour — YVOIRE contour injection into the anteromedial malar region

SUMMARY:
This study is purposed to evaluate the long-term efficacy and safety of repeat treatment of YVOIRE contour injected into the anteromedial malar region in subjects who have completed the LG-HACL014 study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects who have completed the LG-HACL014 study
* Have anteromedial malar region volume loss at least a one-point worse on the MFAS compared with 2 weeks after treatment in the LG-HACL014 study
* Accept the obligation not to receive any other mid facial procedures or treatments during the study
* Signed informed consent
* Those who fall under one of the following 3 cases

  1. Males or females who are surgically sterile
  2. Post-Menopausal females who are above 45 years of age and 2 years after the last menstruation
  3. Fertile premenopausal females or males without having a surgical sterilization, who have agreed to use at least two contraception methods (one of the barrier methods must be included) for up to 14 days after the repeat treatment of the investigational device to avoid pregnancy

Exclusion Criteria:

* Have a history of hypertrophic scars or keloids
* Other criteria as identified in the protocol

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Mid Face Aesthetic Scale (MFAS) score | 2, 26, and 52 weeks after repeat treatment
  Mean of MFAS score as assessed by the independent blinded rater

SECONDARY OUTCOMES:
Mid Face Aesthetic Scale (MFAS) score | 2, 26, and 52 weeks after repeat treatment
  Changes of MFAS score as assessed by the independent blinded rater
Mid Face Aesthetic Scale (MFAS) Responder rate | 2, 26, and 52 weeks after repeat treatment
  MFAS Responder (at least a one-point improvement on the MFAS) rate as assessed by the independent blinded rater
Global Aesthetic Improvement Scale (GAIS) score | 2, 26, and 52 weeks after repeat treatment
  Mean of GAIS score as assessed by subject
Global Aesthetic Improvement Scale (GAIS) Responder rate | 2, 26, and 52 weeks after repeat treatment
  GAIS Responder (at least a one-point improvement on the GAIS) rate as assessed by subject

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea